CLINICAL TRIAL: NCT05179681
Title: Nasal High -Flow Oxygen Therapy Improves Body Temperature Preservation in Non-intubated Thoracoscopic Surgery
Brief Title: High-Flow Oxygen Preserve Intraoperative Body Temperature
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801005RINB
Record Dates: First submitted 2018-01-25; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2018-01

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with non-intubated thoracic surgery
  Interventions: Other: Nasal High -Flow Oxygen Therapy

INTERVENTIONS:
Other: Nasal High -Flow Oxygen Therapy — patients receiving transnasal humidified rapid-insufflation ventilatory exchange

SUMMARY:
Background: Hypothermia would increase the risk of bleeding, infection, cardiac complications and delay recovery. The transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) could not only provide the larger oxygen preserve but also humidified high flow. However, Objectives: We wanted to investigated whether the humidified high flow of THRIVE would affect perioperative body temperature (BT).

Patients and methods: We reviewed the medical records of adult patients undergoing non-intubated video-assisted thoracic surgery (NIVATS) have been retrospective reviewed. All patients have received force air warming. Multiple linear regression analysis was used to determine which factors were associated with BT loss.

Expected result: In patients receiving NIVATS under force air warming, the use of THRIVE may provide more efficiently BT preserve, although the patients with oxygen mask could have acceptable BT preservation. The more BT loss is associated with the advanced age and higher BMI level. The anesthetic duration is not associated with the BT loss.

DETAILED DESCRIPTION:
The goal:In this retrospective study, we aimed to investigate that patients undergoing NIVATS with the use of the THRIVE have better BT than these patients without use the THRIVE.

Methods

A. Study Subjects:

In this retrospective study, the adult patients undergoing nonintubated video-assisted thoracic surgery (NIVATS) with a planned mask or transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) were retrospectively reviewed for patients from the beginning of 2016 to the end of 2017.

Inclusion criteria:

1.Patients who will receive scheduled NOVATS surgery under general anesthesia Patients who met the following criteria were considered candidates for NIVATS: tumours smaller than 6 cm, peripheral lesions, no evidence of severe adhesion, no evidence of chest wall, diaphragm, or main bronchus involvement.

Exclusion criteria:

1.Patients who had potential or confirmed airway complications such as bronchial tumor or hemothorax, morbid obesity (body mass index [BMI] greater than 35), coagulopathy, anatomical deformity or an American Society of Anesthesiology (ASA) classification greater than 3 were excluded.

B. Study Protocol The adult patients undergoing nonintubated video-assisted thoracic surgery (NIVATS) with a planned mask or transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) were retrospectively reviewed for patients from March 2016 to June 2017. All surgical procedures were performed by a single thoracic surgical team using identical clinical protocols, care patterns and perioperative orders. Demographic data and operation outcomes were obtained from the patients' chart review. The core body temperature data, including the last body temperature in the ward before sending to the OR and the first body temperature in the post-anaesthesia care unit (PACU), was obtained from the online records.

C. Methods:

Patients in the mask and thrive groups were all warmed during the whole perioperative periods (beginning in the patients into the operative room (OR) until discharge from OR) using the 3M™ Bair Hugger™ Normothermia System to cover the patients' upper bodies. The temperature of intravenous fluids were kept around 18。C. Below 35。C was selected to define hypothermia because it has been well accepted in the literature as being physiologically significant.

Patients' tympanic temperature as the core temperature was measured on the ward, just before induction and in the OR, and in the postoperative anesthesia unit. For temperature measurements, an infrared tympanic ear thermometer (BRAUN ThermoScan Pro 4000' Welch Allyn, Skaneateles Falls, NY) was used.

Statistical Analysis Categorical data were analysed using the chi-square test. Numerical data were presented as means ± standard deviation unless otherwise specified. Student's t-test was performed to compare the sample means in two independent groups. Paired t-test was performed to compare preoperative and postoperative body temperature change in the THRIVE and mask groups.

Stepwise multivariate linear regression was performed to determine the independent effect of difference body temperature between preoperative and postoperative periods. Variables were included in the model. Age, BMI, using THRIVE or not, intravenous fluid during the operative period, anesthetic duration, and potential confounding factors, which are differed between two groups, were analyzed. A separate stepwise linear regression was performed including patients in the THRIVE and mask groups. A p value < 0.05 was deemed signiﬁcant. Statistical analysis was performed using SPSS 17 statistical software (SPSS, Inc., Chicago, IL, USA).

Study endpoints and sample size calculation The difference between the preoperative and postoperative temperature measurements was compared.

Sample size for the primary outcome end point was determined using the G-power 3 statistical package. Given the SD of core body temperature is around 0.4。C in the general surgical population, a moderate effect size corresponds to a mean temperature difference of 0.2。C between groups. There were 212 patients needed.

ELIGIBILITY:
Inclusion Criteria:

1.Patients who will receive scheduled NOVATS surgery under general anesthesia Patients who met the following criteria were considered candidates for NIVATS: tumours smaller than 6 cm, peripheral lesions, no evidence of severe adhesion, no evidence of chest wall, diaphragm, or main bronchus involvement.

Exclusion Criteria:1. Patients who had potential or confirmed airway complications such as bronchial tumor or hemothorax, morbid obesity (body mass index [BMI] greater than 35 kg·m-2), coagulopathy, anatomical deformity or an American Society of Anesthesiology (ASA) classification greater than 3 were excluded.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing nonintubated video-assisted thoracic surgery (NIVATS) with either a facemask or transnasal humidified rapid-insufflation ventilatory exchange (THRIVE)
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
body temperature changes | before operations, and arrival at postoperative care unit
  the differences of body temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Ya-Jung, Cheng, Taipei, Taiwan